CLINICAL TRIAL: NCT00652587
Title: A Randomized Controlled Trial of Hepatectomy With Adjuvant Transcatheter Arterial Chemoembolization Versus Hepatectomy Alone for Stage IIIA Hepatocellular Carcinoma
Brief Title: Hepatectomy With or Without Transcatheter Arterial Chemoembolization for Stage IIIA Hepatocellular Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Ministry of Health, China (Other Government)
Responsible Party: Cancer Center, Sun Yat-sen University, Cancer Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC_001
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-03

CONDITIONS: Hepatocellular Carcinoma; Hepatectomy; Chemoembolization
Keywords: hepatocellular carcinoma; hepatectomy; chemoembolization; randomized controlled trial; prognosis
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Hepatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A, LRTACE (Experimental): hepatectomy with adjuvant transcatheter arterial chemoembolization
  Interventions: Procedure: hepatectomy and transcatheter arterial chemoembolization
- B, LR (Active Comparator): hepatectomy alone
  Interventions: Procedure: hepatectomy

INTERVENTIONS:
Procedure: hepatectomy and transcatheter arterial chemoembolization — partial hepatectomy with adjuvant transcatheter arterial chemoembolization
  Arms: A, LRTACE
Procedure: hepatectomy — hepatectomy alone
  Other Names: hepatectomy alone
  Arms: B, LR

SUMMARY:
The purpose of this study is to evaluate whether hepatectomy combining with adjuvant transcatheter arterial chemoembolization (TACE) for Stage IIIA hepatocellular carcinoma (HCC) resulting better long-term survival outcome when compared with hepatectomy alone.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the most common malignancies in the world, and the prevalence is increasing in the United States. Hepatectomy is still considered as the potentially curative treatment for HCC. Unfortunately, long-term survival after hepatectomy is still unsatisfactory because of the high incidence of tumor recurrence, especially intrahepatic recurrence.

Stage IIIA hepatocellular carcinoma (HCC) include multiple tumors more than 5 cm or tumor involving a major branch of the portal or hepatic vein(s) in the International Union Against Cancer (UICC) TNM staging for liver tumors, sixth edition 2002. Until now there are controversies in the management of Stage IIIA HCC. According to the Barcelona -Clinic-Liver-Cancer (BCLC) proposal, Stage IIIA HCC represented as intermediate or advanced disease. The European Association for Study of the Liver (EASL) and the American Association for the Study of Liver Diseases (AASLD) recommended randomized controlled trials of chemoembolization or new agents for such stage of disease. Whereas in Asian areas, such as China or Japan, partial hepatectomy or reductive surgery (with or without adjuvant therapy) was performed for multiple advanced HCC or tumor with a major branch of the portal or hepatic vein(s) invasion, although no prospective study to assess the therapeutic efficacy and safety. On the other hand, transcatheter arterial chemoembolization (TACE) is the most widely used primary treatment for unresectable HCC. It was also used as the optional treatment of relapsed disease. However, the efficacy of TACE used as adjuvant therapy following hepatectomy remains controversial. Neither are there large randomized controlled trials to address this field. Therefore, a randomized controlled trial was performed in our cancer center to compare hepatectomy with adjuvant TACE and hepatectomy alone for the Stage IIIA HCC.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients > 18 years and <=70 years of age
* Patients who have an ECOG PS of 0 or 1.
* a preoperative diagnosis of HCC with no previous treatment;
* compensated cirrhosis with Child-Pugh class A, B or no cirrhosis;
* multiple tumors more than 5 cm or tumor involving a major branch of the portal or hepatic vein(s) on preoperative investigations, and on intraoperative ultrasound and gross examination of the liver during the surgery;
* on exploration and intraoperative ultrasound the tumor could safely be resected without grossly remaining tumors, and the patient was judged to have adequate liver functional reserve to survive the operation.

Exclusion Criteria:

* Patient compliance is poor
* Previous or concurrent cancer that is distinct in primary site or histology from HCC, EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis & T1). Any cancer curatively treated > 3 years prior to entry is permitted.
* History of cardiac disease:

  * congestive heart failure > New York Heart Association (NYHA) class 2;
  * active coronary artery disease (myocardial infarction more than 6 months prior to study entry is permitted);
  * cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers, calcium channel blocker or digoxin; or
  * uncontrolled hypertension (failure of diastolic blood pressure to fall below 90 mmHg, despite the use of 3 antihypertensive drugs).
* Active clinically serious infections (> grade 2 National Cancer Institute [NCI]-Common Terminology Criteria for Adverse Events [CTCAE] version 3.0)
* Known history of human immunodeficiency virus (HIV) infection
* Known Central Nervous System tumors including metastatic brain disease
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry
* Distantly extrahepatic metastasis
* History of organ allograft
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Known or suspected allergy to the investigational agent or any agent given in association with this trial
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within seven days prior to the start of study drug. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial.
* Excluded therapies and medications, previous and concomitant:

  * Prior use of any systemic anti-cancer treatment for HCC, eg. chemotherapy, immunotherapy or hormonal therapy (except that hormonal therapy for supportive care is permitted). Antiviral treatment is allowed, however interferon therapy must be stopped at least 4 weeks prior randomization.
  * Prior use of systemic investigational agents for HCC
  * Autologous bone marrow transplant or stem cell rescue within four months of start of study drug

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2002-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
overall survival rates | 1-, 3-, and 5-year

CONTACTS AND LOCATIONS:
Overall Officials: GUO Rong-ping, MD, Principal Investigator — Department of Hepatobilliary Surgery, Cancer Center, Sun Yat-sen University
Locations (1):
- Department of Hepatobilliary Surgery, Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Edwards BK, Brown ML, Wingo PA, Howe HL, Ward E, Ries LA, Schrag D, Jamison PM, Jemal A, Wu XC, Friedman C, Harlan L, Warren J, Anderson RN, Pickle LW. Annual report to the nation on the status of cancer, 1975-2002, featuring population-based trends in cancer treatment. J Natl Cancer Inst. 2005 Oct 5;97(19):1407-27. doi: 10.1093/jnci/dji289. PMID 16204691
- [Background] Lopez PM, Villanueva A, Llovet JM. Systematic review: evidence-based management of hepatocellular carcinoma--an updated analysis of randomized controlled trials. Aliment Pharmacol Ther. 2006 Jun 1;23(11):1535-47. doi: 10.1111/j.1365-2036.2006.02932.x. PMID 16696801
- [Background] Fattovich G, Stroffolini T, Zagni I, Donato F. Hepatocellular carcinoma in cirrhosis: incidence and risk factors. Gastroenterology. 2004 Nov;127(5 Suppl 1):S35-50. doi: 10.1053/j.gastro.2004.09.014. PMID 15508101
- [Background] Llovet JM, Bru C, Bruix J. Prognosis of hepatocellular carcinoma: the BCLC staging classification. Semin Liver Dis. 1999;19(3):329-38. doi: 10.1055/s-2007-1007122. PMID 10518312
- [Background] Bruix J, Sherman M; Practice Guidelines Committee, American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma. Hepatology. 2005 Nov;42(5):1208-36. doi: 10.1002/hep.20933. No abstract available. PMID 16250051
- [Background] Ku Y, Iwasaki T, Tominaga M, Fukumoto T, Takahashi T, Kido M, Ogata S, Takahashi M, Kuroda Y, Matsumoto S, Obara H. Reductive surgery plus percutaneous isolated hepatic perfusion for multiple advanced hepatocellular carcinoma. Ann Surg. 2004 Jan;239(1):53-60. doi: 10.1097/01.sla.0000103133.03688.3d. PMID 14685100
- [Background] Fan J, Zhou J, Wu ZQ, Qiu SJ, Wang XY, Shi YH, Tang ZY. Efficacy of different treatment strategies for hepatocellular carcinoma with portal vein tumor thrombosis. World J Gastroenterol. 2005 Feb 28;11(8):1215-9. doi: 10.3748/wjg.v11.i8.1215. PMID 15754408